CLINICAL TRIAL: NCT03492489
Title: An Open-Label, Expanded Access Protocol of Cemiplimab in Patients With Metastatic or Locally Advanced Cutaneous Squamous Cell Carcinoma Who Are Not Candidates for Surgery
Brief Title: Expanded Access Protocol for Cemiplimab in Metastatic or Locally Advanced Cutaneous Squamous Cell Carcinoma
Status: No longer available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R2810-ONC-17103
Record Dates: First submitted 2018-03-30; First posted 2018-04-10 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Cutaneous Squamous Cell Carcinoma
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: cemiplimab — Intravenous (IV) administration
  Other Names: REGN2810

SUMMARY:
The objective of this program is to provide access to cemiplimab (REGN2810) to patients with metastatic cutaneous squamous cell carcinoma (mCSCC) or locally advanced cutaneous squamous cell carcinoma (laCSCC) who are not candidates for surgery prior to cemiplimab (REGN2810) being commercially available.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of invasive Cutaneous Squamous Cell Carcinoma (CSCC)
2. Hepatic function:

   1. Total bilirubin ≤1.5 x upper limit of normal (ULN; if liver metastases ≤3 x ULN).
   2. Transaminases ≤3 x ULN (or ≤5.0 x ULN, if liver metastases)
   3. Alkaline phosphatase ≤2.5 x ULN (or ≤5.0 x ULN, if liver or bone metastases) Patients with hepatic metastases: If transaminase levels (AST and/or ALT) are >3 x but ≤5 x ULN, total bilirubin must be ≤1.5 x ULN. If total bilirubin is >1.5 x but ≤3 x ULN, both transaminases (AST and ALT) must be ≤3 x ULN
3. Renal function: serum creatinine ≤1.5 x ULN or estimated creatinine clearance (CrCl) >30 mL/min
4. Bone marrow function:

   1. Hemoglobin ≥9.0 g/dL
   2. Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
   3. Platelet count ≥75 x 10^9/L
5. Patients not candidates for surgery include the examples below, but are not limited to:

   * Metastatic disease (distant or nodal)
   * Recurrence in the same location and curative resection is unlikely
   * Significant local invasion that precludes complete resection
   * Surgery may result in severe disfiguration or dysfunction
   * Other conditions deemed to be contraindicating for surgery

Key Exclusion Criteria:

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs). The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism that required only hormone replacement, or psoriasis that does not require systemic treatment
2. Prior treatment with other immune modulating agents that was (a) within fewer than 4 weeks (28 days) prior to the first dose of cemiplimab (REGN2810), or (b) associated with immune-mediated adverse events (AEs) that were ≥ Grade 1 within 90 days prior to the first dose of cemiplimab (REGN2810), or (c) associated with toxicity that resulted in discontinuation of the immune-modulating agent
3. Continuous immunosuppressive corticosteroid treatment (doses >10 mg prednisone daily or equivalent) within 2 weeks prior to the first dose of cemiplimab (REGN2810)Note: Patients who require brief course of steroids (eg, as prophylaxis for imaging studies) are not excluded
4. Active uncontrolled infection requiring therapy, including infection with human immunodeficiency virus, or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
5. History of pneumonitis within the last 5 years

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Regeneron Pharmaceuticals